CLINICAL TRIAL: NCT06981845
Title: Sirolimus With corTicOsteroid TheraPy for Rapid rEcurrences of Coronary Unexplained In-stent Restenosis (STOP-RECUR) Study
Brief Title: Sirolimus With corTicOsteroid TheraPy for Rapid rEcurrences of Coronary Unexplained In-stent Restenosis
Acronym: STOP-RECUR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Kefei Dou, MD, Professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-2645; 2025-2645 (Other: Fuwai Hospital, China National Center for Cardiovascular Diseases)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: In-stent Restenosis Lesion; Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD))
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction | interventions — Immunosuppression Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppressive therapy group (Experimental): (1) prednisone + sirolimus and (2) standard coronary artery disease therapy
  Interventions: Drug: Immunosuppressive therapy
- placebo control group (Placebo Comparator): (1) placebo and (2) standard coronary artery disease therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Immunosuppressive therapy — prednisone + sirolimus
  Arms: Immunosuppressive therapy group
Drug: Placebo — Placebo
  Arms: placebo control group

SUMMARY:
This study aims to evaluate, through a multicenter, prospective, double-blind, randomized, placebo-controlled clinical trial, whether immunosuppressive therapy improves target lesion-related cardiovascular outcomes compared to placebo treatment in patients with Rapid rEcurrence of Coronary Unexplained in-stent Restenosis (RECUR).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Able to understand the trial design and sign an informed consent form
3. Patients meeting the RECUR definition
4. Satisfactory results from revascularization within the past two weeks
5. Receiving standard secondary prevention medication for coronary heart disease with treatment targets achieved

Exclusion Criteria:

Pregnant women, individuals known to be allergic to the study drug, those currently participating in other interventional clinical trials, or participants deemed unsuitable for this study based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | During the 1 year follow-up
  Time to first occurrence of Target vessel failure (TVF), defined as cardiac death, target vessel-related myocardial infarction, or clinically driven target vessel revascularization.

IPD SHARING:
Plan to Share IPD: No